CLINICAL TRIAL: NCT06843811
Title: A Pilot Phase 2 Study With Long-Term Extension to Assess the Safety and Efficacy of Sirolimus in Patients With Leigh Syndrome Caused by Genetically-Confirmed Mitochondrial Respiratory Chain Deficiency
Brief Title: Sirolimus for Leigh Syndrome
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Matthew Demczko (Other)
Responsible Party: Sponsor-Investigator, Matthew Demczko, Sponsor-Investigator, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-022433
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Leigh Syndrome
MeSH Terms: conditions — Leigh Disease | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 2A (Experimental): Participants will receive Sirolimus for at least 24 weeks at a starting dose of 0.8 to 1.3 mg/m2 two (2) times daily.
  Interventions: Drug: Sirolimus
- Long-Term Extension (Experimental): Eligible participants may continue Sirolimus treatment for up to two (2) years.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Sirolimus will be given at a starting dose of 0.8 to 1.3 mg/m2 twice daily, depending on subject age and weight.
  Other Names: Rapamune; Rapamycin

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the drug Sirolimus in participants with Leigh syndrome.

DETAILED DESCRIPTION:
This is a pilot phase 2 study with long-term extension to evaluate the safety and efficacy of enteral sirolimus in patients with genetically-confirmed Leigh syndrome.

Sirolimus will be given daily at a starting dose of 0.8 to 1.3 mg/m2 depending on subject age, weight, and BSA (body surface area). Dosage will be adjusted as needed based on sirolimus trough level to maintain patients within a range of 5 to10 ng/mL, a level lower than what is targeted in renal transplant recipients. Patients will be followed through this study for up to 24 weeks in the active phase. Participants who are eligible for the long-term extension may choose to stay on drug for up to 2 years thereafter

ELIGIBILITY:
Inclusion Criteria:

1. Genetically-confirmed diagnosis of Leigh syndrome with neurodevelopmental manifestations, which include documented developmental delay, developmental regression, or abnormal neurologic exam findings including but not limited to hypotonia, hypertonia, dystonia, chorea, nystagmus, ataxia, dysmetria, tremor or muscle weakness.
2. Age 6 months to 55 years at the time of enrollment.
3. Weight ≥ 5 kg at the time of enrollment.
4. Adequate liver function as evidenced by total bilirubin < 1.5x upper limit of normal (ULN) and liver function tests, alanine transaminase (ALT) and aspartate aminotransferase (AST), < 3x ULN.
5. Adequate renal function as evidenced by glomerular filtration rate (GFR) > 60 mL/min/1.73m2 (cystatin C for pediatric population).
6. Normal hematologic parameters as defined as:

   1. Absolute neutrophil count (ANC) ≥ 1.0 x 109/L
   2. Platelet count ≥ 100,000/mm3 (100 x 109/L)
   3. Hemoglobin ≥ 9 g/dL
7. Non-fasting serum triglycerides and cholesterol < 300 mg/dL.
8. Serum amylase and lipase < 2x ULN.
9. Adequate immunoglobulin levels as outlined below that, in the opinion of the investigator, will not place the patient at increased risk of infection.

   1. Immunoglobulin G (IgG) ≥ 200 mg/dL
   2. Immunoglobulin M (IgM) ≥ 30 mg/dL
   3. Immunoglobulin A (IgA) ≥ 10 mg/dL
10. All sexually active participants must agree to use effective contraception:

    1. Females of child-bearing potential must agree to use effective contraception without interruption from 28 days prior to starting Investigational Product (IP) throughout 3 months after last dose of IP and have a negative urine pregnancy test result at screening and agree to ongoing pregnancy testing during the course of the study.
    2. Male patients must practice abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study and throughout 3 months after the last dose of investigational drug.
11. The patient or parent(s)/legal guardian(s) is/are willing and able to comply with the study visit schedule and other protocol requirements, in the opinion of the investigator.
12. The patient or the patient's parent(s)/legal guardian(s) understand(s) and voluntarily sign(s) the informed consent documents(s) prior to any study-related assessments/procedures being conducted.

Exclusion Criteria:

1. Cardiac ejection fraction ≤ 50 %, shortening fraction ≤ 25% on cardiac echocardiogram within one year of screening and/or severe end-organ hypo-perfusion syndrome (secondary to cardiac failure) resulting in lactic acidosis.
2. Patients with implanted cardiac assist/medical devices (including pacemakers), unless device was implanted prophylactically, and the patient is clinically asymptomatic.
3. In the opinion of the investigator, clinically significant ECG and/or echocardiogram alterations at the time of screening.
4. Myocardial infarction within 6 months prior to enrollment.
5. Symptomatic congestive heart failure (CHF), unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension, or unstable coronary artery disease.
6. Prior history of hypersensitivity to sirolimus or other mTOR (Mechanistic Target of Rapamycin inhibitors).
7. Prior history of angioedema requiring treatment or cessation of a presumed causative agent.
8. Planned surgical procedure during the study period.
9. Confirmed or highly suspected immunodeficiency disorder(s), including but not limited to, common variable immune deficiency (CVID), complement deficiency, etc.
10. Clinically significant proteinuria that requires ongoing medical therapy.
11. Any uncontrolled psychiatric or medical condition which, in the opinion of the investigator, would interfere with the patient's participation in the study.
12. Patients who are breastfeeding or are pregnant.
13. History of solid organ transplant (kidney, liver, heart, lung) or bone marrow transplant.
14. Treatment with any investigational drug (i.e., a drug for which there is no approved indication), including an investigational drug for mitochondrial disease within 1 month prior to receiving the first dose of study drug (or within 3 months for a trial with an investigational biologic).
15. Patients with confirmed or suspected increased intracranial pressure, pseudotumor cerebri (PTC)/idiopathic intracranial hypertension, and or papilledema.
16. Currently active malignancy (other than adequately treated non-melanoma skin cancers [i.e., squamous cell and/or basal cell carcinoma], carcinoma in situ of the cervix, or other adequately treated carcinoma in situ) and/or ongoing treatment for malignancy are ineligible. Patients are not considered to have a currently active malignancy if they have completed therapy and are free of disease for ≥ 1 year.
17. Recent infection requiring systemic anti-infective treatment that was completed ≤ 14 days prior to enrollment.
18. Uncontrolled diabetes mellitus, as defined by HbA1c > 8%, despite adequate therapy.
19. History of interstitial lung disease and/or pneumonitis.
20. Use of strong inhibitors and/or inducers of cytochrome P450 (CYP) 3A4 (CYP3A4) and/or p-glycoprotein (p-GP) within the 14 days prior to receiving the first dose of study drug. Additionally, use of any known CYP3A4 substrates with a narrow therapeutic window (e.g., fentanyl, alfentanil, astemizole, cisapride, dihydroergotamine, pimozide, quinidine, terfenadine) within the 14 days prior to receiving the first dose of study drug.
21. Use of medications with a high risk of angioedema
22. Known human immunodeficiency virus (HIV), active hepatitis B or hepatitis C infection(s).

Ages: 6 Months to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Rate of Adverse Events | Up to 2.5 years
  Adverse events will be measured according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE). Incidence of AEs will be reported.
Rate of Intercurrent Infection and Hospitalization | Up to 2.5 years
  Each infection and hospitalization will be reported.
Incidence of abnormal safety lab values | Up to 2.5 years
  Count of clinically significant changes from baseline in safety labs
Sirolimus Trough Level | Up to 2.5 years
  Measure of Sirolimus level in the blood. Sirolimus dosage will be adjusted as needed in order to maintain a sirolimus trough level within a range of 5 to 10 ng/mL. The number of out-of-range results will be reported.

SECONDARY OUTCOMES:
Change in MM-COAST Score | Baseline up to end of study (up to 2.5 years)
  Mitochondrial Myopathy-Composite Assessment Tool (MM-COAST) is a composite assessment tool used to measure the domains of muscle strength, muscle fatigue, balance, dexterity, and exercise intolerance.
  Scores are assigned for each domain assessment, based on z-score or % decrement for muscle fatigue, summed and averaged to achieve a domain score. The mean domain score is reported as the MM-COAST Composite Score.
Change in GMFM (Gross Motor Function Measure) Score | Baseline up to end of study (up to 2.5 years)
  The GMFM is a clinical tool used assess changes in gross motor functions in 5 dimensions (1. lying and rolling, 2. sitting, 3. crawling and kneeling, 4. standing, and 5. walking, running, and jumping). Each task is scored as 0-does not initiate, 1-initiates, 2-partially completes, and 3-completed.
  Item scores are summed to calculate raw and percent scores for each of the five dimensions. Dimension percent scores are averaged to obtain an overall total score.
Change in Movement Disorder-Childhood Rating Score (MDCRS) | Baseline up to end of study (up to 2.5 years)
  The MDCRS is a scale used to evaluate the impact of movement disorder on patient motor function and daily living activities. Severity of movement disorder in different regions of the body at rest, and during specific tasks, is ranked from 0 (no movement disorder) to 4 (severe movement disorder).
  Item scores are summed to calculate total score, with a higher total score indicating greater overall impact of movement disorder on daily functioning.
CGI Scale | Baseline up to end of study (up to 2.5 years)
  The CGI (Clinical Global Impression Scale) is a 3-item clinician-rated scale used to assess severity of illness, global improvement, and therapeutic response. Degree of global improvement for participants receiving sirolimus will be assessed by the investigator and rated on a scale 7-point scale based on improvement from baseline from 1 (very much improved) to 7 (very much worse). A lower score indicates greater response to treatment.
Change in Barry-Albright Dystonia Scale (BADS) | Baseline up to end of study (up to 2.5 years)
  The Barry-Albright Dystonia Scale is used to assess dystonia in 8 bodily regions: eyes, mouth, neck, trunk, and each upper and lower extremity. Each bodily region is scored based on a scale from 0 (absent) to 4 (severe symptoms). Total BADS score ranges from 0 (dystonia absent) to 32 (severe dystonia).
Change in Scale for the Assessment and Rating of Ataxia (SARA) | Baseline up to end of study (up to 2.5 years)
  The SARA is an 8-item performance-based scale that assesses ataxia. Patients are evaluated based on their ability to perform a series of tasks with a cumulative score ranging from 0 (no ataxia) to 40 (most severe ataxia).
Newcastle Pediatric Mitochondrial Disease Scale (NPMDS) | Baseline up to end of study (up to 2.5 years)
  The NPMDS evaluates the progression of mitochondrial disease in pediatric patients in 4 domains: current function, system specific involvement, current clinical assessment and quality of life. Domain scores are summed for total score with higher scores indicating worse conditions.
Newcastle Adult Mitochondrial Disease Scale (NMDAS) | Baseline up to end of study (up to 2.5 years)
  Evaluation of disease progression in adults. Each question in the NMDAS section I-III has a possible score from 0-5. The total score is calculated by summing the scores obtained for each question. The higher the score the more severe the disease.
Change in PEDI-CAT Score | Baseline up to end of study (up to 2.5 years)
  Pediatric Evaluation of Disability Inventory Computer Adaptive Test (PEDI-CAT) is a test that evaluates daily functional activities. A t-score of 50 represents the function of the general population (SD of 10). A t-score below 30 reflects poor performance compared to the general population.
  The range for the scores are 20-80.
Patient Global Impression of Change (PGIC) | Baseline up to end of study (up to 2.5 years)
  Patients rate their impression of overall change from baseline on a 7-point scale from 0 (no change or condition is worse) to 7 (a great deal better). PGIC indicates a patient's belief of treatment efficacy
Change in PedsQL | Baseline up to end of study (up to 2.5 years)
  Pediatric Quality of Life Inventory (PedsQL) is a 23-item questionnaire that evaluates health-related quality of life that is reported as 3 summary scores including Physical Health, Psychosocial Health and School/Work, as well as a total score (sum of summary scores). Total score ranges from 0-100 with a higher score indicating better quality of life.
Change in Karnofsky-Lansky | Baseline up to end of study (up to 2.5 years)
  Karnofsky Lansky Scale: 0-100. 0-40: Unable to care for self, requires equivalent of institutional or hospital care; disease may be progressing rapidly. 50-70: Unable to work; able to live at home and care for most personal needs; varying amount of assistance needed. 80-100: Able to carry on normal activity and to work; no special care needed.
Change in MFIS | Baseline up to end of study (up to 2.5 years)
  The MFIS (Modified Fatigue Impact Scale) evaluates fatigue using a total MFIS score (0-84), where higher scores indicate greater impact of fatigue on an individual's activities and scores above 38 are considered to be indicative of fatigue.
  The MFIS is calculated from the sum of three subscales: the Physical Subscale (0-36), the Cognitive Subscale (0-40), and the Psychosocial Subscale (0-8), where higher scores indicate a greater impact of fatigue in each domain.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Demczko, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson SC, Yanos ME, Kayser EB, Quintana A, Sangesland M, Castanza A, Uhde L, Hui J, Wall VZ, Gagnidze A, Oh K, Wasko BM, Ramos FJ, Palmiter RD, Rabinovitch PS, Morgan PG, Sedensky MM, Kaeberlein M. mTOR inhibition alleviates mitochondrial disease in a mouse model of Leigh syndrome. Science. 2013 Dec 20;342(6165):1524-8. doi: 10.1126/science.1244360. Epub 2013 Nov 14. PMID 24231806
- [Background] Johnson SC, Yanos ME, Bitto A, Castanza A, Gagnidze A, Gonzalez B, Gupta K, Hui J, Jarvie C, Johnson BM, Letexier N, McCanta L, Sangesland M, Tamis O, Uhde L, Van Den Ende A, Rabinovitch PS, Suh Y, Kaeberlein M. Dose-dependent effects of mTOR inhibition on weight and mitochondrial disease in mice. Front Genet. 2015 Jul 22;6:247. doi: 10.3389/fgene.2015.00247. eCollection 2015. PMID 26257774
- [Background] Tinker RJ, Falk MJ, Goldstein A, George-Sankoh I, Xiao R, Adang L, Ganetzky R. Early developmental delay in Leigh syndrome spectrum disorders is associated with poor clinical prognosis. Mol Genet Metab. 2022 Apr;135(4):342-349. doi: 10.1016/j.ymgme.2022.02.006. Epub 2022 Feb 19. PMID 35216885
- [Background] Zheng X, Boyer L, Jin M, Kim Y, Fan W, Bardy C, Berggren T, Evans RM, Gage FH, Hunter T. Alleviation of neuronal energy deficiency by mTOR inhibition as a treatment for mitochondria-related neurodegeneration. Elife. 2016 Mar 23;5:e13378. doi: 10.7554/eLife.13378. PMID 27008180